CLINICAL TRIAL: NCT00899132
Title: The Role of TAB3 Protein in Tumorigenesis
Brief Title: Studying a Tumor Marker for Testicular Cancer, Skin Cancer, Small Intestine Cancer, and Pancreatic Cancer
Status: Terminated | Type: Observational
Why Stopped: Study due for continuing review
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CASE5Y06; P30CA043703 (NIH); CASE5Y06 (Other: Case Comprehensive Cancer Center); CASE-5Y06-CC191 (Other: Cancer Center IRB)
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2015-09-29 (Estimated); Status verified 2015-09

CONDITIONS: Non-melanomatous Skin Cancer; Pancreatic Cancer; Small Intestine Cancer; Testicular Germ Cell Tumor
Keywords: skin cancer; small intestine cancer; pancreatic cancer; malignant testicular germ cell tumor; testicular teratoma
MeSH Terms: conditions — Pancreatic Neoplasms; Testicular Germ Cell Tumor; Skin Neoplasms; Testicular Neoplasms; Teratoma, Testicular | interventions — In Situ Hybridization; Immunologic Techniques

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Tumor tissue samples from paraffin-embedded tissue blocks.
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: in situ hybridization — Tumor tissue samples from paraffin-embedded tissue blocks are analyzed for TAB3 transcript and protein expression using in situ hybridization and immunostaining with TAB3 cRNA probe and antibody. Antibodies against the proteins involved in the NFkB signaling pathway (e.g., p65, TAK1, MyD88, and Akt) are used in the immunostaining assays.
Genetic: protein expression analysis — Tumor tissue samples from paraffin-embedded tissue blocks are analyzed for TAB3 transcript and protein expression using in situ hybridization and immunostaining with TAB3 cRNA probe and antibody. Antibodies against the proteins involved in the NFkB signaling pathway (e.g., p65, TAK1, MyD88, and Akt) are used in the immunostaining assays.
Other: immunologic technique — Tumor tissue samples from paraffin-embedded tissue blocks are analyzed for TAB3 transcript and protein expression using in situ hybridization and immunostaining with TAB3 cRNA probe and antibody. Antibodies against the proteins involved in the NFkB signaling pathway (e.g., p65, TAK1, MyD88, and Akt) are used in the immunostaining assays.

SUMMARY:
RATIONALE: Studying samples of tumor tissue from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer.

PURPOSE: This research study is evaluating a tumor marker for testicular cancer, skin cancer, small intestine cancer, and pancreatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To identify TAB3 transcript/protein as a molecular marker of cancer, specifically testicular, skin, small intestine, and pancreatic cancer.
* To characterize TAB3 and its signaling networks that are involved in tumorigenesis.

OUTLINE: Tumor tissue samples from paraffin-embedded tissue blocks are analyzed for TAB3 transcript and protein expression using in situ hybridization and immunostaining with TAB3 cRNA probe and antibody. Antibodies against the proteins involved in the NFkB signaling pathway (e.g., p65, TAK1, MyD88, and Akt) are used in the immunostaining assays.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Paraffin tissue blocks from surgical pathology cancer cases, specifically testicular, skin, small intestine, and pancreatic cancer, available

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Primary care center
Sampling Method: Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2007-02; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Identification of TAB3 transcript/protein as a molecular marker of cancer | end of study
Characterization of TAB3 and its signaling networks that are involved in tumorigenesis | end of study

CONTACTS AND LOCATIONS:
Overall Officials: Ge Jin, PhD, Study Chair — Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center
Locations (1):
- Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States